CLINICAL TRIAL: NCT01416402
Title: A Phase 2, Open-label Study to Evaluate the Safety and Efficacy of Arhalofenate (MBX-102) in Combination With Febuxostat for the Treatment of Hyperuricemia in Patients With Gout
Brief Title: Open Label Safety/Efficacy Study of Arhalofenate in Combination With Febuxostat for Hyperuricemia in Gout Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M102-21124
Record Dates: First submitted 2011-08-11; First posted 2011-08-15 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Hyperuricemia; Gout
Keywords: Hyperuricemia; gout; serum uric acid
MeSH Terms: conditions — Hyperuricemia; Gout | interventions — arhalofenate; Febuxostat; Colchicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arhalofenate with febuxostat and colchicine (Other)
  Interventions: Drug: Arhalofenate; Drug: Febuxostat; Drug: Colchicine

INTERVENTIONS:
Drug: Arhalofenate — 400 mg once daily orally for two weeks then up-titrated to 600 mg once daily orally for an additional two weeks
  Other Names: MBX-102
Drug: Febuxostat — 80 mg once daily orally for 5 weeks
  Other Names: Uloric
Drug: Colchicine — Colchicine 0.6 mg daily as prophylaxis to prevent gout flares
  Other Names: Colcrys

SUMMARY:
The purpose of this study is to determine whether arhalofenate is safe and effective when dosed in combination with febuxostat in lowering serum uric acid in patients with gout.

ELIGIBILITY:
Inclusion Criteria:

1. Known gout patient (per criteria of the American Rheumatism Association for the classification of the acute arthritis of primary gout in Appendix 3) with a serum uric acid value of at least 8.0 mg/dL at Screening Visit. Patients on allopurinol must agree to discontinue their existing therapy at Visit 1 through the entire duration of the study and must have a sUA value of at least 8.0 mg/dL after a minimum 2 week wash-out at Visit 2.
2. Male or female, 18-75 years of age at Screening Visit
3. All female patients must be surgically sterile or post-menopausal (at least 45 years of age with no history of menses for at least 2 years; or any age with no history of menses for at least 6 months and serum FSH ≥ 40 mIU/mL) or must agree to use two medically accepted methods of contraception including a barrier method (see the list in Appendix 4) for the entire duration of the study unless report of complete sexual abstinence.
4. Female patients must not be pregnant or lactating
5. Male patients with a female partner of child-bearing potential must agree to use condom or the partner must use a medically acceptable method of contraception for the entire duration of the study.
6. Estimated CrCl ≥ 50 mL/min as calculated by the by Cockcroft-Gault method
7. Serum creatinine value must be ≤ 1.3 mg/dL in females and ≤ 1.4 mg/dL in males
8. Patients must have liver function tests (LFTs) ≤ 1.5X ULN for AST, ALT and T-bilirubin, ≤ 2X ULN for ALP, ≤ 3X ULN for GGT; CK ≤ 3X ULN
9. All other clinical laboratory parameters must be within normal limits or considered not clinically significant
10. Electrocardiogram (ECG) must be normal, or if abnormal, considered not clinically significant
11. Patients must have a systolic blood pressure ≤ 160 mm Hg and a diastolic blood pressure ≤ 95 mm Hg; known hypertensive patients controlled with medication other than diuretics (BP reading as above) may be included
12. Patients must agree to remain in-clinic for 37 days consecutively and agree to follow the study procedures as described in the protocol

Exclusion Criteria:

1. Treatment with any ULT other than allopurinol (e.g., probenecid, benzbromarone, febuxostat, or pegloticase) within two weeks of the Screening Visit
2. Known or suspected secondary hyperuricemia (e.g. due to myeloproliferative disorder, or organ transplant).
3. Diagnosis of xanthinuria
4. History of documented or suspected kidney stones
5. Known infection with the human immunodeficiency virus (HIV) or history of viral hepatitis type B or C
6. History of illicit drug or alcohol abuse within one year of Screening Visit
7. History of significant pulmonary disease, upper gastrointestinal (GI) bleeding, documented peptic ulcer disease (unless known H. pylori infection treated successfully without recurrence), or nephrotic syndrome within three years of Screening Visit
8. History of stroke, TIA, acute myocardial infarction (MI), congestive heart failure (CHF) (NYHA Class II-IV), angina pectoris, coronary intervention procedure (including but not limited to angioplasty, stent placement, coronary revascularization), lower extremity bypass procedure, systemic or intracoronary fibrinolytic therapy within 5 years of screening
9. Malignancy within five years of Screening Visit (except successfully treated basal cell carcinoma)
10. Body mass index (BMI) > 42 kg/m2
11. Current or expected requirement for anticoagulant therapy [except for low-dose (≤ 325 mg/day) aspirin and/or Plavix® 75 mg/day]
12. Rheumatoid arthritis or other autoimmune disease requiring ongoing treatment
13. Current or expected treatment with potent CYP3A4 inhibitors (See Appendix 6), cytotoxic agents (azathioprine, mercaptopurine, cyclosporine, cyclophosphamide, etc.), ranolazine, digoxin, theophyline, desipramine, sulphonylurea, thiazolidinedione, diuretics, atypical antipsychotic agents, or phenytoin
14. Chronic treatment with non-steroidal anti-inflammatory drugs (NSAIDs use to treat acute gout flares is permitted)
15. Current or expected treatment with systemic corticosteroids (except topical, ophthalmic, intra-articular, or inhaled at a dose < 1600 μg/day) other than to treat acute gout flares
16. Known hypersensitivity to colchicine or febuxostat
17. Treatment with any other investigational therapy within the 30 days prior to the Screening Visit, or patients who received at least one dose of blinded study medication while enrolled in any previous arhalofenate trial
18. Any other condition that compromises the ability of the patient to provide informed consent or to comply with the objectives and procedures of this protocol, as judged by the investigator and/or medical monitor

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving sUA <6.0 mg/dL, <5.0 mg/dL, <4.0 mg/dL and <3.0 mg/dL at the end of combination treatment period with each of the doses of arhalofenate | 36 days

CONTACTS AND LOCATIONS:
Locations (1):
- Overland Park, Kansas, United States